CLINICAL TRIAL: NCT06100198
Title: Evaluation of the Effect of Nutrition and Exercise Program Intervention on the Health of Community-dwelling Older Adults
Brief Title: The Effect of Nutrition and Exercise Program on the Health of Community-dwelling Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TCHIRB-11206012-E
Record Dates: First submitted 2023-10-17; First posted 2023-10-25 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Healthy Aging; Nutrition, Healthy; Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior | interventions — Nutritional Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): A one-group pretest-posttest design was adopted. Participants participated in 3 nutrition and exercise courses, each lasting 2 hours (including 1 hour nutrition course and 1 hour exercise course) with an interval of 1 week between each course. All subjects underwent anthropometric measurements and completed questionnaires one week before the start of the course and one week after the end of the course. A repeat assessment was conducted 6 months after the course intervention.
  Interventions: Other: nutrition and exercise program

INTERVENTIONS:
Other: nutrition and exercise program — Nutrition courses include understanding malnutrition and sarcopenia; understanding the six major food categories and their requirements; and understanding protein-rich food sources. Exercise courses include understanding exercise types, flexibility exercises, and muscle strength training exercises.

SUMMARY:
The purpose of this study is to design a nutrition and exercise course for the elderly adults in the community, and to evaluate the effectiveness of this course intervention on the nutritional knowledge, nutritional status, sarcopenia, and health status of the elderly in the community. This study adopted convenience sampling and targeted 108 community elders over 65 years old in Taipei City. All participants receive 3 nutrition and exercise courses. Each course was separated by one week. Measurements and collections were conducted one week before and one week after the course. BMI (body mass index), muscle mass, calf circumference, grip strength, Mini Nutritional Assessment Form Short Form (MNA-SF), SARC-F scale, Taiwan Short Form 36 Health Scale (SF-36) and nutrition knowledge and attitude and behavioral questionnaires will be collected to evaluate the effectiveness of the course.

DETAILED DESCRIPTION:
The elderly population in Taiwan, aged over 65, has exceeded 14%, officially marking the country's transition into an aging society. This demographic shift has brought forth numerous health-related challenges among the elderly, including malnutrition, sarcopenia, and frailty, thereby increasing the risk of falls, cognitive dysfunction, and morbidity rates. This also results in rising disability and mortality rates, ultimately driving up healthcare costs.

The primary aim of this study is to develop a nutrition and exercise program for elderly individuals within the community. This program will be carried out in collaboration with a team of nutrition and exercise professionals. Furthermore, the study seeks to assess the effectiveness of this intervention on the nutritional awareness, nutritional status, sarcopenia, and overall health of elderly community members.

The study employed convenience sampling and included 108 community elders aged over 65 from Taipei City, all of whom were sourced from the community congregated meal stations. Each participant received three nutrition and exercise courses, with each course separated by a week. Measurements for body weight, BMI (body mass index), muscle mass, calf circumference, grip strength, Mini Nutritional Assessment Form Short Form (MNA-SF), SARC-F scale, Taiwan Short Form 36 Health Scale (SF-36), as well as pre- and post-course knowledge, attitude, and behavior assessments were conducted one week before and after the program.

After collecting the questionnaire data, SPSS version 22 (IBM Corp., Armonk, NY, USA) was used for data storage and statistical analysis. A p-value less than 0.05 was considered statistically significant. Descriptive statistical analysis methods, including mean, standard deviation, and percentages, were employed to provide a basic overview of the participant group. To understand differences and correlations between variables, the study utilized Chi-square and Paired Sample T-test methods.

Through this project, the investigators aim to evaluate the impact of the nutrition and exercise course intervention for elderly individuals in Taipei City. This endeavor will empower participants to incorporate nutrition and exercise strategies into daily lives, ultimately fostering better health outcomes for the elderly adults.

ELIGIBILITY:
Inclusion Criteria:

1. Citizens aged 65 and above, residing in communities in Taipei City.
2. Clear consciousness and the ability to communicate in Mandarin and Taiwanese.
3. Capability to move freely.

Exclusion Criteria:

1. Individuals with cognitive impairment who are unable to cooperate with the measurements.
2. Those unable to walk.
3. Individuals with obvious edema of the lower limbs.
4. Those with hand disabilities (such as fractures, arthritis, or stroke) preventing the measurement of grip strength.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | One week before the first class, one week after the third class, and 6 months after the course intervention.
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters.
Calf circumference | One week before the first class, one week after the third class, and 6 months after the course intervention.
  The widest part of the calf was measured with a non-elastic tape applied flat on the skin and parallel to the floor.
Hand grip strength | One week before the first class, one week after the third class, and 6 months after the course intervention.
  Grip strength is measured using a hand-held dynamometer (TTM-YD, Tsutsumi Industries, Tokyo, Japan）.
Muscle mass | One week before the first class, one week after the third class, and 6 months after the course intervention.
  Muscle mass is measured using a Inbody H20B Smart Full Body Composition Analyzer Scale.
Nutritional status | One week before the first class, one week after the third class, and 6 months after the course intervention.
  Nutritional status was assessed using the Mini Nutritional Assessment Form Short Form (MNA-SF), a six-item instrument with scores ranging from 0 to 14 points. A total score of MNA-SF <8, 8-11, and >11 indicates malnutrition, risk of malnutrition, and no malnutrition, respectively.
The risk of sarcopenia | One week before the first class, one week after the third class, and 6 months after the course intervention.
  Strength, assistance with walking, rising from a chair, climbing stairs, and falls (SARC-F) questionnaire scores. The SARC-F scores range from 0 (best) to 10 (worst). Patients with a total score ≥4 were considered to be at risk of sarcopenia.
Taiwan Short 36 Health Scale (SF-36) | One week before the first class, one week after the third class, and 6 months after the course intervention.
  The SF-36 is a self-rated scale consisting of 36 items that assess health-related quality of life (HRQoL) in eight health dimensions. This questionnaire consists of 36 questions, focusing on the following two norm-based composite scales: physical component scale (PCS) and mental component scale (MCS). The PCS includes four subscales: physical functioning (PF), role functioning due to limitations in physical problems (RP), bodily pain (BP), and general health (GH). The MCS also includes four subscales: vitality (VT), social functioning (SF), role limitations due to emotional problems (RE), and mental health (MH). The subscales are reported as scores that range from 0 to 100. Higher scores indicate more favourable levels of function.
Nutritional knowledge, attitudes, and behaviors | One week before the first class, one week after the third class, and 6 months after the course intervention.
  Using a self-administered questionnaire to study the relationships among dietary knowledge, attitudes, and behaviors. The scores range from 0 to 20, 0 to 12, 0 to 9 for nutritional knowledge, attitudes, and behaviors respectively. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ping Chang, Doctor, Principal Investigator — Taipei City Hospital
Locations (1):
- Huanyu International Culture and Education Foundation Guting Branch, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No